CLINICAL TRIAL: NCT04048811
Title: A Multi-Center, Randomized, Open-Label, Positive-Controlled Phase II Clinical Trial Evaluating the Efficacy and Safety of HSK3486 Injectable Emulsion for Induction and Maintenance of General Anesthesia in Elective Surgery Patients.
Brief Title: A Clinical Trial Evaluating the Efficacy and Safety of HSK3486 Injectable Emulsion in Elective Surgery Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486-204
Record Dates: First submitted 2019-07-31; First posted 2019-08-07 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Induction and Maintenance of General Anesthesia
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Masking Description: Upon enrollment of the 40 subjects, 6 more subjects will be enrolled by West China Hospital of Sichuan University. These 6 subjects will not be randomized, but will directly enter into propofol induction + HSK3486 maintenance group for study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK3486 (Experimental): HSK3486 induction + maintenance group
  Interventions: Drug: HSK3486
- Propofol (Active Comparator): Propofol induction + maintenance group
  Interventions: Drug: Propofol
- Propofol HSK3486 (Other): Propofol induction + HSK3486 maintenance group
  Interventions: Drug: Propofol HSK3486

INTERVENTIONS:
Drug: HSK3486 — The induction dose is 0.4mg/mg. The initial maintenance dose of the first 6 subjects is 1 mg/kg/h. For the subsequent enrolled subjects, the investigator could adjust the subsequent initial maintenance dose according to the dose response of the first 6 subjects, so as to explore the optimal initial maintenance dose. The range of the initial maintenance dose is 1 (± 0.5) mg/kg/h, i.e. the minimum initial maintenance dose should not be less than 0.5 mg/kg/h, and the maximum should not be more than 1.5 mg/kg/h.
  Arms: HSK3486
Drug: Propofol — The induction dose is 2.0mg/mg. The initial maintenance dose of the first 2 subject is 5 mg/kg/h. For the subsequent enrolled subjects, the investigator could adjust the subsequent initial maintenance dose according to the dose response of the first 2 subjects, so as to explore the optimal initial maintenance dose. The adjustment range of the initial maintenance dose is 5 (± 2.5) mg/kg/h, i.e. the minimum initial maintenance dose should not be less than 2.5 mg/kg/h, and the maximum should not be more than 7.5 mg/kg/h.
  Arms: Propofol
Drug: Propofol HSK3486 — The induction dose of Propofol is 2.0mg/mgThe initial maintenance dose of HSK3486 is fixed at 1 mg/kg/h, without adjustment.
  Arms: Propofol HSK3486

SUMMARY:
This is a multi-center, randomized, open-label, positive-controlled (propofol) phase II clinical trial. The study plans to enroll approximately 46 eligible subjects. Among them, 40 subjects will be randomly assigned to HSK3486 treatment group (30 cases) and propofol control group (10 cases) in a ratio of 3:1. The subjects will be enrolled competitively at all study sites. Upon enrollment of the 40 subjects, 6 more subjects will be enrolled by West China Hospital of Sichuan University. These 6 subjects will not be randomized, but will directly enter into propofol induction + HSK3486 maintenance group for study.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients requiring tracheal intubation under general anesthesia and a non-emergent, non-cardiothoracic, non-extracerebral, and non-nasal endoscopic elective surgery for an estimated duration of about 1-6 h, with an bleeding volume of ≤ 1000 mL
2. Aged ≥ 18 and ≤ 65 years old, regardless of gender;
3. American Society of Anesthesiologists (ASA) Class I-III;
4. Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2;
5. The vital signs during the screening period meet the following criteria:

   * Respiratory rate ≥ 10 and ≤ 24 breaths/min;
   * Blood oxygen saturation (SpO2) ≥ 95% when inhaling;
   * Systolic blood pressure (SBP) ≥ 90 mmHg and ≤ 160 mmHg;
   * Diastolic blood pressure (DBP) ≥ 60 mmHg and ≤ 100 mmHg;
   * Heart rate ≥ 55 beats/min and ≤ 100 beats/min;
6. The laboratory parameters measured at screening period reach the following criteria:

   * Neutrophil count ≥ 1.5 × 109/L;
   * Platelet count ≥ 80 × 109/L;
   * Hemoglobin ≥ 90 g/L (no blood transfusion within 14 days);
   * ALT and AST ≤ 3.0 × upper limit of normal (ULN);
   * Total bilirubin ≤ 1.5 × ULN;
   * Serum creatinine ≤ 1.5 × ULN.
7. Subjects who understand the procedures and methods of this study, and are willing to complete the trial in strict accordance with clinical trial protocol and sign the informed consent.

Exclusion Criteria:

1. Patients with contraindications to general anesthesia or previous history of anesthesia accidents;
2. Known hypersensitivity to excipients and ingredients found in propofol injection and HSK3486 injectable emulsion (soybean oil, glycerin, triglycerides, egg lecithin, sodium oleate, and sodium hydroxide), benzodiazepines, opioids, rocuronium bromide, and sugammadex sodium; cross-reactivity to halogenated anesthetics, jaundice or unexplained fever from previous use of halogenated anesthetics; contraindications to propofol;
3. Medical history or evidence of any of the following prior to screening, which may increase sedation/anesthesia risk:

   * History of cardiovascular disease: Uncontrolled hypertension or SBP > 160 mmHg and/or DBP > 100 mmHg despite antihypertensive treatment, severe arrhythmia, heart failure, Adams-Stokes syndrome, unstable angina, myocardial infarction occurring in almost 6 months prior to screening, and history of tachycardia/bradycardia requiring medication, third-degree atrioventricular block or QTcF ≥ 450 ms (male) or ≥ 470 ms (female) (corrected using Fridericia's formula) during screening period.
   * Respiratory system disorders: Respiratory insufficiency, history of bronchospasm requiring treatment within 3 months prior to screening, acute respiratory tract infection with obvious symptoms such as fever, wheezing, or productive cough within 1 week prior to administration of the study drug;
   * History of craniocerebral disease: Patient with a history of craniocerebral injury, convulsions, epilepsy, intracranial hypertension, cerebral aneurysm, or cerebrovascular accident; history of schizophrenia, mania, chronic use of antipsychotics, or cognitive impairment.
   * Gastrointestinal disease history: Gastrointestinal retention, active hemorrhage, or circumstances that may lead to reflux and aspiration.
   * Diabetic patients with uncontrolled blood glucose (fasting blood glucose ≥ 11.1 mmol/L, and/or random blood glucose ≥ 13.6 mmol/L).
   * Patients with a history of uncontrolled and clinically significant liver, kidney, blood system, nervous system or metabolic system diseases judged by the investigator to be unsuitable for this trial.
   * History of alcohol abuse within 3 months prior to screening, where alcohol abuse refers to daily alcohol drinking > 2 units of alcohol (1 unit = 360 mL of beer or 45 mL of liquor with 40% alcohol or 150 mL of wine).
   * History of drug abuse within 3 months prior to screening.
   * Serious infection, trauma, or major surgery within 4 weeks prior to screening.
4. Any one of the following respiratory risks before/during screening:

   * Asthma history, and stridor.
   * Sleep apnea syndrome.
   * History of malignant hyperthermia or family history.
   * History of failed tracheal intubation.
   * Judged by the investigator to have difficult airway or judged as difficult tracheal intubation (modified Mallampati score III or IV);
5. Received any of the following drugs or therapies prior to screening:

   * Participated in other drug trials within 1 month prior to screening.
   * Using the drugs that may affect QT interval within 2 weeks prior to screening.
   * Using propofol, other sedatives/anesthetics, and/or opioid analgesics or compounds containing analgesics within 3 days prior to screening.
6. Women who are pregnant or breastfeeding; women of child-bearing potential or men who are unwilling to use contraception during the trial; Subjects who are planning pregnancy within 1 month after the completion of the trial (including male subjects);
7. Subjects judged by the investigator to be unsuitable for participating in this trial for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-05-23 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Success rate of anesthesia maintenance | During maintenance of general anesthesia on day 1
  During the maintenance of anesthesia, the subject is not recovered and no remedial anesthetic is used
Number of patients with adverse events | Pre-dose to 48 hours post-dose
  Safety endpoints

SECONDARY OUTCOMES:
Success rate of anesthesia induction | During induction of general anesthesia on day 1
  During the induction of anesthesia, the subject achieves successful induction (i.e., MOAA/S ≤ 1) after administration of the study drug (up to 2 additional doses), and no remedial anesthetic is used.
Success rate of anesthesia | During induction and maintenance of general anesthesia on day 1
  The proportion of subjects who are successfully induced and successfully maintain anesthesia in all subjects.
Changes in Bispectral index | During maintenance of general anesthesia on day 1
  Bispectral index (BIS) is used to adjust the administration dose during anesthesia maintenance to maintain BIS at 40-60
Time to successful induction of anesthesia | Time to successful induction of anesthesia on day 1
  A period of time from the start of the first administration of the study drug to the first time when MOAA/S is ≤ 1.
Time to recovery from anesthesia | A period of time from discontinuation of the study drug to recovery after the end of surgery on day 1.
  6.Record the time when MOAA/S = 5 is reached for the first time.
Time to respiratory recovery | A period of time from discontinuation of the study drug to respiratory recovery after the end of surgery on day 1.
  Respiratory rate ≥ 8 breaths/min and the tidal volume ≥ 5 mL/kg.
Time to extubation | A period of time from discontinuation of the study drug to extubation after the end of surgery on day 1.
Time to leaving the operating room | A period of time from discontinuation of the study drug to leaving the operating room after the end of surgery on day 1.
Time to leaving postanesthesia care unit(PACU) | A period of time from discontinuation of the study drug to leaving PACU after the end of surgery on day 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China